CLINICAL TRIAL: NCT02343146
Title: Healthy Eating, Physical Activity, and Glycemic Control in Young Children With T1D
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Randi Streisand (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor-Investigator, Randi Streisand, MD, Children's National Research Institute
Organization: Children's National Research Institute (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 5649; DP3DK103998 (NIH)
Record Dates: First submitted 2015-01-08; First posted 2015-01-21 (Estimated); Last update posted 2019-08-02 (Actual); Status verified 2019-08

CONDITIONS: Diabetes Mellitus, Type 1
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Type One Training (TOT) (Experimental): The intervention group will receive the proposed intervention composed of peer parent consultants, telephone and in-person sessions with a trained interventionist, and SMS text messaging aimed at improving child glycemic control through improved nutrition and physical activity.
  Interventions: Behavioral: Type One Training (TOT)
- Comparison (No Intervention): The comparison group will receive usual care with the diabetes team.

INTERVENTIONS:
Behavioral: Type One Training (TOT) — The intervention is comprised of a number of modes of delivery including in person, use of parent peer consultant, telephone intervention, and text messaging. The intervention is based on Social Cognitive Theory and previous work of the investigators.The focus of the intervention is on working with parents to improve child eating and physical activity behaviors as a means of improving glycemic control in very young children with type 1 diabetes.
  Arms: Type One Training (TOT)

SUMMARY:
The incidence of type 1 diabetes (T1D) in young children (age <5 years) is rising. The burden of responsibility for disease management rests on parents and caregivers to check blood sugar, administer insulin, and monitor diet and physical activity to maintain tight glycemic control. This occurs at a vulnerable time in life when children's behavior is unpredictable, their T1D is difficult to control, and parenting stress is elevated. Despite behavioral interventions that have demonstrated success in reducing rates of parent stress and improving child behavior, improvements in young children's glycemic control has not been sufficiently achieved. The investigators' research will attempt to achieve this goal through the development and pilot of an innovative behavioral intervention for T1D in parents of young children. The focus of the intervention is on improving young children's nutrition and physical activity through the use of parent consultants and delivery of intervention through phone and text messaging. The study will be conducted in two phases. In Phase 1, 10 primary caregivers of young children (<5 years) diagnosed with T1D for at least 6 months will receive the intervention and then be assessed at 3- and 6- months post baseline on indices of behavior and glycemic control (including continuous glucose monitoring). Participants will also complete in-depth surveys to provide qualitative as well as quantitative data. At the end of Phase 1, the data will be analyzed and used to develop the intervention further for Phase 2. During Phase 2, 60 participants and their children will be randomized to either the revised intervention (treatment) or usual care (control) condition. Intervention components include: T1D management support delivered by trained lay parent consultants, and T1D parenting strategies specific to improving eating and physical activity behaviors delivered by bachelor's level behavioral assistants via telephone and text messaging. Biomedical and psychosocial measurements (including HbA1c, physical activity, nutrition, mealtime behavior, parenting stress, quality of life) will occur at baseline and 3- and 6-months post baseline. The results of this work will ultimately lead to a program which can improve young children's T1D management and glycemic control that can be translated into a variety of clinical practice settings.

DETAILED DESCRIPTION:
Young children (<5 years) comprise a growing number of persons diagnosed with type 1 diabetes (T1D)--a costly, chronic illness [1, 2]. Early age at diagnosis and poor glycemic control during these early years increases risk for development of serious diabetes-related complications (ref). Thus, these years represent a critical period for establishing proper patterns of T1D management and glycemic control in young children [7]. In addition to young children's daily reliance on parents for T1D care, such as blood glucose (BG) monitoring and insulin administration, careful attention must be paid to diet and physical activity regulation. Behavioral interventions supporting and enhancing T1D management among parents of these young children have the potential for significant impact on children's glycemic control as well as developmentally important outcomes, and may reduce both immediate and long-term clinical and public health burdens of T1D complications.

Although multicomponent behavioral interventions for parents of young children with T1D demonstrate potentially promising psychosocial outcomes [8-10], concomitant improvements in children's glycemic control from these interventions remain elusive. Two critical areas not yet addressed directly in interventions is the promotion of healthy eating and engagement in consistent physical activity in young children, nor the behavioral strategies to support parents in these challenges that occur multiple times daily (e.g., each meal/snack, each physical activity experience). The current proposal utilizes the extensive expertise of our multidisciplinary team to refine and pilot an innovative and translatable intervention targeting eating and physical activity behaviors directly associated with glycemic control in young children that can ultimately be adopted outside of research settings. The investigators' prior successful clinical research efforts engaging parents of young children with T1D in behavioral interventions (R01 DK080102) places them in a unique position to further design and pilot this intervention and ultimately be well poised to run a future full-scale efficacy trial.

The current proposal shifts the investigators' prior interventions' focus away from parental stress and instead highlights behavioral strategies promoting healthy eating and engagement in consistent physical activity, as well as nutrition and physical activity links to glycemic control. Based upon positive preliminary data the investigators will utilize novel assessment (accelerometry, personal activity monitors (PAM), and continuous glucose monitors (CGM)) and intervention components (parent consultants and trained intervention telephone counselors), with the intervention being delivered via telephone and in-person. The investigators will follow an iterative mixed methods approach to refine the intervention from Phase 1 to Phase 2. During phase 1 the investigators will pre-pilot the intervention by examining feasibility and acceptability in 10 parents (of children ages 1-5 yrs with a minimum of 1 yr duration of diabetes). The investigators will use qualitative interviews, questionnaire, and objective (CGM, accelerometry) data to help refine key intervention components and discern best areas for intervention target (i.e., low glycemic breakfast or different meal; planned physical activity or increasing steps through daily living; PAM or accelerometry). This phase will include soliciting feedback from the advisory board leading to further refinement of the intervention and manual of procedures. During phase 2 the investigators will execute a pilot randomized trial evaluating whether glycemic control and developmentally-important outcomes (child feeding and physical activity) in young children with T1D can be favorably impacted. Phase 2 will include 60 parents (of children ages 1-5 yrs) randomly allocated to either the intervention (n=30) or standard care (n=30). Assessments will be completed 3 times (T1, T2-immediately post intervention, and T3-6 months post-intervention). Clinical, biological, and behavioral diabetes outcomes will be measured. Specific Aims for this trial are:

Aim 1. Pilot test and refine innovative and feasible assessment and intervention components for T1D control in young children, and examine acceptability and impact in parents of young children. At the conclusion of Phase 1, this Aim results in an innovative intervention program, supported by state of the art assessment tools and preliminary data. The investigators hypothesize that the intervention will be associated with high feasibility and acceptability, improved T1D management, and reduction of behavioral challenges related to eating and physical activity.

Aim 2. Determine the intervention's efficacy for improving young children's glycemic control and parent's management of eating and physical activity behaviors. The investigators hypothesize that the Phase 2 pilot will demonstrate that relative to usual care, the intervention will evidence 1) Significantly better glycemic control (i.e., HbA1c <8.5% and higher percentage of BG levels in the 100-200 mg/dl range, per ADA recommendations) and 2) Significantly fewer child feeding and activity behavior problems (e.g., food refusal, dawdling at mealtimes, physical inactivity). 3. Mediating effects of eating and physical activity on glycemic control will also be explored.

Aim 3. Explore the feasibility of program implementation in a larger scale efficacy trial, and in clinical T1D management. Using a purposeful sample subset of parents in the intervention condition, the investigators will use qualitative interviews to further examine the impact of the intervention, and assist in further refinement prior to a larger scale trial. The investigators will also interview advisory board members including members of the health care team to gather system- and provider-level data about key capacities to inform the integration of our intervention into patient/work flow in anticipation of a larger efficacy trial.

ELIGIBILITY:
Inclusion Criteria:

* parent of a child age 1-5 and their target child (children are considered secondary participants)
* child with a minimum of 1 year duration of T1D
* parents must have ready and consistent access to a mobile telephone with text messaging capability

Exclusion Criteria:

* Parent participants cannot have serious mental illness or developmental disability that would limit participation
* Child participants cannot have other life-threatening disease (e.g., cancer, cystic fibrosis) or developmental disability (e.g., autism, mental retardation)
* Parent participants must be able to adequately understand, speak, and read English

Ages: 21 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2015-12 (Actual); Primary Completion 2019-05 (Actual); Study Completion 2019-08 (Actual)

PRIMARY OUTCOMES:
Glycemic Control/HbA1c | 6 months post intervention
  Change in glycemic control from baseline to 6 months post intervention

SECONDARY OUTCOMES:
Child eating as measured by Remote Food Photography by the parent | 6 months post intervention
  Change in child eating behaviors from baseline to 6 months post intervention

CONTACTS AND LOCATIONS:
Overall Officials: Randi Stresiand, PhD, Principal Investigator — Children's National Research Institute
Locations (1):
- Children's Research Institute, Washington D.C., District of Columbia, United States

REFERENCES:
- [Derived] Mackey ER, Tully C, Rose M, Hamburger S, Wang J, Herrera N, Cogen F, Henderson C, Monaghan M, Hornack S, Streisand R. Promoting glycemic control in young children with type I diabetes: Results from a pilot intervention for parents. Fam Syst Health. 2022 Jun;40(2):239-251. doi: 10.1037/fsh0000672. PMID 35666897